CLINICAL TRIAL: NCT02250469
Title: A Randomised Pilot Study to Assess differenCes in tHe Subjects' Experience of stimulAtion-Induced paRaesthesiA Between Two Different Spinal Cord sTimulation dEvices: the Axium® DoRsal Root Ganglion Stimulation System Versus the Prime Advanced Dorsal Column Stimulation System
Brief Title: A Randomised Pilot Study to Assess Differences in Stimulation Induced Paresthesia Between 2 Spinal Cord Stimulation Systems
Acronym: CHARACTER SCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-SMI-2014
Record Dates: First submitted 2014-09-09; First posted 2014-09-26 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axium SCS System (Active Comparator): Implantation with the Axium Neurostimulator
  Interventions: Device: Treatment with the Axium SCS system
- Medtronic SCS System (Active Comparator): Implantation with the Medtronic Prime Advanced Dorsal Column Stimulation System
  Interventions: Device: Treatment with the Medtronic SCS System

INTERVENTIONS:
Device: Treatment with the Axium SCS system
  Arms: Axium SCS System
Device: Treatment with the Medtronic SCS System
  Arms: Medtronic SCS System

SUMMARY:
12-SMI-2014 is a post-market, randomised, pilot study to identify and rate differences in patient experiences with two different types of Spinal Cord Stimulator devices which are routinely used to treat chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is appropriate for SCS implantation according to standard criteria
2. Subject is >18 to <75 years old
3. Subject is able and willing to comply with the follow-up schedule and protocol
4. Subject has chronic (> 6 months) uni/bi-lateral neuropathic pain in the lower limb(s) (below the knee) with predominant foot pain
5. Minimum baseline pain rating of 50 mm on the VAS in the primary region of pain
6. Subject is able to provide written informed consent

Exclusion Criteria:

1. Subject has no other exclusion criteria for SCS implantation according to standard criteria
2. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
3. Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
4. Subject has participated in another clinical study within 30 days
5. Subject has been previously treated with and failed to respond to an implantable neuromodulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Specificity of Stimulation Induced Paresthesia | 3 Months post implantation
  A comparative analysis will be made between groups to determine the percentage of a patients painful and non-painful anatomy that is covered by stimulation induced paresthesia
Stability of Stimulation Induced Paresthesia | 3 Months post implantation
  A comparative analysis will be made between groups to determine any changes in the intensity of stimulation induced paresthesia in response to changes in body position
Patient Interactions with System | 3 Months post implantation
  A comparative analysis will be made between groups to determine the number of device interactions patients need to have on average, daily

CONTACTS AND LOCATIONS:
Overall Officials: M W Hollmann, Prof, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academisch Medisch Centrum, Amsterdam, Netherlands